CLINICAL TRIAL: NCT00726986
Title: Phase II Trial of Sorafenib in Conjunction With Chemotherapy and as Maintenance Therapy in Extensive-Stage Small Cell Lung Cancer
Brief Title: Sorafenib, Cisplatin, and Etoposide in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Extreme toxicity
Sponsor: Afshin Dowlati, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Afshin Dowlati, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE8507; P30CA043703 (NIH); CASE8507 (Other: Case Comprehensive Cancer Center); CASE-8507-CC486 (Other: Cancer Center IRB)
Record Dates: First submitted 2008-07-31; First posted 2008-08-01 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Etoposide; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib, Cisplatin, and Etoposide (Experimental)
  Interventions: Drug: cisplatin; Drug: etoposide; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: cisplatin — Cisplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Drug: etoposide — Etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Drug: sorafenib tosylate — Oral sorafenib tosylate twice daily beginning on day 1 of course 1 and continuing for up to 1 year in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving sorafenib together with cisplatin and etoposide works in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the 1-year progression-free survival of patients with extensive-stage small cell lung cancer treated with sorafenib tosylate in combination with cisplatin and etoposide.
* To evaluate the 1-year overall survival and response rate in these patients.
* To evaluate the safety of these drugs in these patients.

OUTLINE: This is a multicenter study.

Patients receive cisplatin IV over 30-60 minutes on day 1 and etoposide IV over 60 minutes on days 1-3. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients also receive oral sorafenib tosylate twice daily beginning on day 1 of course 1 and continuing for up to 1 year in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of extensive-stage small cell lung cancer
* No untreated brain metastases

  * No active symptoms related to brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Hemoglobin ≥ 9.0 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver involvement)
* Creatinine ≤ 1.5 times ULN
* INR < 1.5 or PT/PTT normal
* No history of cardiac disease, including any of the following:

  * NYHA class III-IV congestive heart failure
  * Unstable angina (i.e., anginal symptoms at rest)
  * Onset of angina within the past 3 months
  * Myocardial infarction within the past 6 months
* No cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg, despite optimal medical management
* No thrombolic or embolic events, such as cerebrovascular accident or transient ischemic attacks, within the past 6 months
* No pulmonary hemorrhage/bleeding event ≥ CTCAE grade 2 within the past 4 weeks
* No other hemorrhage/bleeding event ≥ CTCAE grade 3 within the past 4 weeks
* No known HIV infection or chronic hepatitis B or C infection
* No active clinically serious infection > CTCAE grade 2
* No serious non-healing wound, ulcer, or bone fracture
* No evidence or history of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 4 weeks
* No known or suspected allergy to sorafenib tosylate or to any other drug given during the study
* No condition that would impair the patient's ability to swallow whole pills
* No known malabsorption problem
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

  * Male patients must use effective contraception during and for ≥ 3 months after completion of sorafenib tosylate

PRIOR CONCURRENT THERAPY:

* Prior radiotherapy to the brain allowed
* No prior chemotherapy
* More than 4 weeks since prior major surgery or open biopsy
* No concurrent Hypericum perforatum (St. John's wort) or rifampin
* Concurrent anti-coagulation treatment, such as warfarin or heparin, allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center; Nathan Pennell, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (11):
- United States (11):
  - Columbia Presbyterian, New York, New York
  - Lake/University Ireland Cancer Center, Cleveland, Ohio
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - CCF-Fairview Hospital, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - UH-Monarch, Mayfield Heights, Ohio
  - UH-Firelands, Sandusky, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 patients were enrolled into the trial from 3 sites between August 2008 and November 2011. Patients were recruited from University Hospitals Case Medical Center and Cleveland Clinic in Cleveland Ohio and Columbia Presbyterian in New York.
Groups:
- Sorafenib, Cisplatin, and Etoposide: Sorafenib, Cisplatin, and Etoposide for 4 cycles (months) during maintenance phase. If no disease progression continue with sorafenib for a maximum of 12 months.
Period: Induction Phase
Arm/Group | Sorafenib, Cisplatin, and Etoposide
Started | 18
Maintance | 3
Completed | 3
Not Completed | 15
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 2
Not completed — Death | 2
Not completed — Lack of Efficacy | 5
Not completed — Secondary Disease | 2
Period: Maintenance Phase
Arm/Group | Sorafenib, Cisplatin, and Etoposide
Started | 3
Completed | 0
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib, Cisplatin, and Etoposide
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival(PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever comes first.
Time Frame: 1-year
Population: Patients who received at least one dose of the study drug were considered evaluable for both toxicity and response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib, Cisplatin, and Etoposide
Number analyzed (Participants) | 16
months | 5.1 [1.2 to 8.2]

2. Secondary Outcome: Median Overall Survival
Description: Overall survival is measured from the date of chemotherapy treatment (date of cycle 1 of induction chemotherapy) until death and censored at the date of last follow-up for survivors.
Time Frame: 1-year
Population: Patients who received at least one dose of the study drug were considered evaluable for both toxicity and response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib, Cisplatin, and Etoposide
Number analyzed (Participants) | 16
months | 7.4 [2.5 to 10.2]

3. Secondary Outcome: Response Rate
Description: The Response Evaluation Criteria in Solid Tumors (RECIST) were used to assess response to the treatment.
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: reevaluated for response every 8 weeks
Population: Patients who received at least one dose of the study drug were considered evaluable for both toxicity and response.
Measure: Number; unit: participants
Arm/Group | Sorafenib, Cisplatin, and Etoposide
Number analyzed (Participants) | 17
participants
  Complete Response (CR) | 1
  Partial Response (PR) | 7
  Stable Disease (SD) | 1
  Progressive Disease (PD) | 8

4. Secondary Outcome: Safety
Description: Number of patients that experienced grade 3-4-5 treatment related toxicities. Toxicity was graded by the National Cancer Institute Common Terminology Criteria version 3.0.
Time Frame: Treatment repeats every 21 days for 4 courses in the absence of unacceptable toxicity.
Population: Patients who received at least one dose of the study drug were considered evaluable for both toxicity and response.
Measure: Number; unit: participants
Arm/Group | Sorafenib, Cisplatin, and Etoposide
Number analyzed (Participants) | 17
participants | 14

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events while on treatment and post-treatment follow up for up to 1 year.
Arm/Group | Sorafenib, Cisplatin, and Etoposide
Serious Adverse Events (participants affected / at risk) | 14/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib, Cisplatin, and Etoposide (N=17)
Creatinine (Investigations) | 1
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1
Hemorrhage, GI (Gastrointestinal disorders) | 2
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3
Peripheral arterial ischemia (Vascular disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Renal/Genitourinary- Glomerular Filtration Rate (Renal and urinary disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 2
Renal/Genitourinary (Renal and urinary disorders) | 2
Pain, Oral Cavity (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Dizziness (General disorders) | 1
Thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib, Cisplatin, and Etoposide (N=17)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 8
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4
Cardiac Arrhythmia (Cardiac disorders) | 4
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 6
Distension/bloating, abdominal (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Edema-limbs (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 11
Flatulence (Gastrointestinal disorders) | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 8
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 10
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 9
Hot flashes/flushes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 3
Insomnia (Psychiatric disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 7
Mood alteration - Anxiety (Psychiatric disorders) | 2
Mood alteration - Depression (Psychiatric disorders) | 3
Mucositis/stomatitis - Oral cavity (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 10
Neuropathy: sensory (Nervous system disorders) | 4
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 10
PTT (Partial Thromboplastin Time) (Investigations) | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 4
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 3
Pain - Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 3
Pain - Extremity-limb (Metabolism and nutrition disorders) | 2
Pain - Head/headache (Nervous system disorders) | 6
Pain - Pelvis (General disorders) | 2
Platelets (Blood and lymphatic system disorders) | 8
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2
Rigors/chills (General disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7
Taste alteration (dysgeusia) (Nervous system disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 2
Vision-blurred vision (Eye disorders) | 2
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 5
Weight loss (Investigations) | 5
Creatinine (Metabolism and nutrition disorders) | 2
Phosphate (Metabolism and nutrition disorders) | 2
Infection (Infections and infestations) | 3

LIMITATIONS AND CAVEATS:
This study was terminated after enrolling 18 patients on the basis of excessive toxicity observed and preliminary efficacy data showing that study was unlikely to meet primary end point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes